CLINICAL TRIAL: NCT01682460
Title: Pilot Study on the Use of Artificial Tears to Treat Dry Eye in Glaucoma Patients
Acronym: IVES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18262
Record Dates: First submitted 2012-08-29; First posted 2012-09-11 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Glaucoma; Dry Eyes
MeSH Terms: conditions — Glaucoma; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Refresh Tears Lubricant Eye Drops (Allergan) (Experimental): Artificial tears eye drops QID for 1 month
  Interventions: Drug: Refresh Tears Lubricant Eye Drops (Allergan)

INTERVENTIONS:
Drug: Refresh Tears Lubricant Eye Drops (Allergan) — Eye drops QID for 1 month

SUMMARY:
Research indicates that many people who are being treated for glaucoma have dry eyes. The purpose of this study is to test the use of artificial tears to alleviate dryness signs and symptoms in people who are using medication to treat glaucoma. The study hypothesis is that the use of artificial tears will result in an improvement in clinical signs and symptoms associated with dry eyes.

ELIGIBILITY:
Inclusion Criteria:

* At least 17 years of age and has full legal capacity to volunteer;
* Has read and signed an information consent letter;
* Is willing and able to follow instructions and maintain the appointment schedule;
* Is a current non-contact lens wearer.
* Has previously been diagnosed with primary open angle glaucoma and is currently being treated with a topical therapeutic agent.
* The glaucoma medication dosage and usage must have been the same for >6 months.
* Shows a minimum score of 2 (sometimes) on the SESOD questionnaire.
* Distance VA of at least 20/40 in each eye with current spectacle correction.

Exclusion Criteria:

* Is participating in any concurrent clinical or research study;
* Has any known active* ocular disease and/or infection; except primary open angle glaucoma.
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
* Is using any systemic or topical medications (with the exception of glaucoma medication) that in the opinion of the investigator may affect a study outcome variable;
* Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
* Is pregnant, lactating or planning a pregnancy at the time of enrolment;
* Has undergone refractive error surgery;
* Is an employee of the Centre for Contact Lens Research;
* Has taken part in another (pharmaceutical) research study within the last 30 days;
* Is currently using artificial tears more than 3 times per day.

  * For the purposes of this study, active ocular disease is defined as infection or inflammation that requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, Principal Investigator — University of Waterloo
Locations (1):
- Centre for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Refresh Tears Lubricant Eye Drops (Allergan)
Started | 15
Completed | 11
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Did not meet inclusion criteria | 2

BASELINE CHARACTERISTICS:
Arm/Group | Refresh Tears Lubricant Eye Drops (Allergan)
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 2
Region of Enrollment [Number; unit: participants]
  Canada | 11

OUTCOME MEASURES:

1. Primary Outcome: Ocular Surface Staining
Description: Corneal staining assessed using slit lamp biomicroscopy on a 1-5 scale where 0=no staining and 5= >30 dots + confluence
Time Frame: At baseline (dispensing visit)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Refresh Tears Lubricant Eye Drops (Allergan)
Number analyzed (Participants) | 11
units on a scale | 1.65 (0.80)

2. Primary Outcome: Ocular Surface Staining
Description: Corneal staining assessed using slit lamp biomicroscopy on a 1-5 scale where 0=no staining and 5= >30 dots + confluence
Time Frame: After 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Refresh Tears Lubricant Eye Drops (Allergan)
Number analyzed (Participants) | 11
units on a scale | 1.55 (0.88)

3. Primary Outcome: Ocular Surface Staining
Description: Corneal staining assessed using slit lamp biomicroscopy on a 1-5 scale where 0=no staining and 5= >30 dots + confluence
Time Frame: After 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Refresh Tears Lubricant Eye Drops (Allergan)
Number analyzed (Participants) | 11
units on a scale | 1.29 (0.89)

4. Primary Outcome: Tear Break up Time With Fluorescein
Description: The time taken for the tear film to break up on the surface of the cornea will be measured using slit lamp biomicroscopy following fluorescein instillation .
Time Frame: At baseline (dispensing visit)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Refresh Tears Lubricant Eye Drops (Allergan)
Number analyzed (Participants) | 11
seconds | 2.88 (2.01)

5. Primary Outcome: Tear Break up Time With Fluorescein
Description: as for outcome 4
Time Frame: After 1 week
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Refresh Tears Lubricant Eye Drops (Allergan)
Number analyzed (Participants) | 11
seconds | 3.41 (2.29)

6. Primary Outcome: Tear Break up Time With Fluorescein
Description: as for outcome 4
Time Frame: After 1 month
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Refresh Tears Lubricant Eye Drops (Allergan)
Number analyzed (Participants) | 11
seconds | 4.01 (2.76)

7. Secondary Outcome: Ocular Surface Disease Index (OSDI) Score
Description: The OSDI is a questionnaire that consists of 12 questions about ocular irritation and the effect of dry eye on vision. For every question, participants check a score between 0 and 4, where 0 equals "none of the time" and 4 equals "all of the time". OSDI scores are calculated according to: OSDI = [(sum of scores for all questions answered)*100] / [(total number of questions answered)*4]. The possible range of the OSDI score is 0 (best possible score) to 100 (worst possible score).
Time Frame: At baseline (dispensing visit)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Refresh Tears Lubricant Eye Drops (Allergan)
Number analyzed (Participants) | 11
units on a scale | 25 (16)

8. Other Pre Specified Outcome: Subjective Ratings of Comfort
Description: Participants completed a standardized grading scale regarding their subjective ratings of comfort (0 = very poor comfort, 100=excellent comfort)
Time Frame: At baseline (dispensing visit)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Refresh Tears Lubricant Eye Drops (Allergan)
Number analyzed (Participants) | 11
units on a scale | 80 (14)

9. Secondary Outcome: Ocular Surface Disease Index (OSDI) Score
Description: as for outcome 7
Time Frame: 1 week after using artificial tears
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Refresh Tears Lubricant Eye Drops (Allergan)
Number analyzed (Participants) | 11
units on a scale | 18 (11)

10. Secondary Outcome: Ocular Surface Disease Index (OSDI) Score
Description: The OSDI is a questionnaire that consists of 12 questions about ocular irritation and the effect of dry eye on vision. For every question, participants check a score between 0 and 4, where 0 equals "none of the time" and 4 equals "all of the time". OSDI scores are calculated according to: OSDI = [(sum of scores for all questions answered)*100] / [(total number of questions answered)*4]. The possible range of the OSDI score is 0 (best possible score) to 100 (worse possible score).
Time Frame: 1 month after using artificial tears
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Refresh Tears Lubricant Eye Drops (Allergan)
Number analyzed (Participants) | 11
units on a scale | 15 (13)

11. Other Pre Specified Outcome: Subjective Ratings of Comfort
Description: Participants completed a standardized grading scale regarding their subjective ratings of comfort (0-100, 0= very poor comfort, 100=excellent comfort)
Time Frame: 1 week after using artificial tears
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Refresh Tears Lubricant Eye Drops (Allergan)
Number analyzed (Participants) | 11
units on a scale | 92 (8)

12. Other Pre Specified Outcome: Subjective Ratings of Comfort
Description: Participants completed a standardized grading scale regarding their subjective ratings of comfort (0-100, 0=very poor comfort, 0 = excellent comfort)
Time Frame: 1 month after using artificial tears
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Refresh Tears Lubricant Eye Drops (Allergan)
Number analyzed (Participants) | 11
units on a scale | 92 (7)

ADVERSE EVENTS:
Arm/Group | Refresh Tears Lubricant Eye Drops (Allergan)
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Refresh Tears Lubricant Eye Drops (Allergan) (N=11)
Corneal marginal keratitis (Eye disorders) | 1 (1) — Unrelated to study drops

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes